CLINICAL TRIAL: NCT02521441
Title: A Multi-center, Randomized, Open-label, Active-controlled, Dose Finding Study to Evaluate the Efficacy and Safety of F-627 Compared to Filgrastim in Women With Breast Cancer Receiving Myelotoxic Chemotherapy.
Brief Title: A Phase II, Dose-finding Study of F-627 in Patients With Breast Cancer Receiving Myelotoxic Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Collaborators: Fudan University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Tongji Hospital (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); RenJi Hospital (Other); Zhejiang Cancer Hospital (Other); Yunnan Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Jiangsu Provincial People's Hospital (Other); Huaxi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-CDR-1-1302
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Neutropenia
Keywords: Neutropenia; Myelotoxic Chemotherapy; G-CSF
MeSH Terms: conditions — Neutropenia | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- F-627, 10 mg/dose (Experimental): F-627 at dose of 10 mg/dose administered by subcutaneous injection on Day 3 of each cycle for up to 4 cycles. EC regimen (Epirubicin and Cyclophosphamide) administered by intravenous injection on Day 1 of each cycle for 4 cycles.
  Interventions: Biological: F-627
- F-627, 20 mg/dose (Experimental): F-627 at dose of 20 mg/dose administered by subcutaneous injection on Day 3 of each cycle for up to 4 cycles. EC regimen (Epirubicin and Cyclophosphamide) administered by intravenous injection on Day 1 of each cycle for 4 cycles.
  Interventions: Biological: F-627
- Filgrastim, 5 mcg/kg/dose (Experimental): Filgrastim of 5 mcg/dose administered by subcutaneous injection for up to two weeks, start from Day 3 of each cycle for up to 4 cycles. EC regimen (Epirubicin and Cyclophosphamide) administered by intravenous injection on Day 1 of each cycle for 4 cycles.
  Interventions: Biological: Filgrastim

INTERVENTIONS:
Biological: F-627 — F-627 at doses of 10 mg/dose or 20 mg/dose, s.c. on Day 3 of each cycle for up to 4 cycles.
  Arms: F-627, 10 mg/dose; F-627, 20 mg/dose
Biological: Filgrastim — Filgrastim at dose of 5 mcg/kg/day for up to 2 weeks, s.c. start from Day 3 of each cycle for up to 4 cycles.
  Other Names: rh G-CSF
  Arms: Filgrastim, 5 mcg/kg/dose

SUMMARY:
This was a randomized, open-label, active-controlled, dose-finding, phase II study to evaluate the efficacy and safety of 2 doses of F-627 compared to Filgrastim in women with breast cancer receiving myelotoxic chemotherapy.

Subjects would be randomized to one of three arms, which were 10 mg/dose of F-627, 20 mg/dose of F-627 or Filgrastim, in an equal ratio.

DETAILED DESCRIPTION:
This phase II study was conducted at 16 clinical centers in China and planned to enroll 150 women with breast cancer who will receive chemotherapy that includes up to 4 cycles of epirubicin and cyclophosphamide, 100 mg/m2 and 600 mg/m2, respectively. Subjects would be randomized to one of three arms, which were 10 mg/dose of F-627, 20 mg/dose of F-627 or Filgrastim, in an equal ratio on Day 1 of the study. Patients will remain on their randomized study drug dose and regimen for each of the following 3 chemotherapy cycles. The chemotherapy to be administered for chemotherapy cycles 2-4 should be the same therapy administered to the subject on Day1.

Chemotherapy will be administrated through intravenous IV) injection on Day 1 of each 21-day cycle and be repeated every 3 weeks for up to four cycles unless a dose delay is necessary. Approximately 48 hours after chemotherapy completion in cycle (day 3 of the cycle), patients will either receive a subcutaneous (SC) injection of F-627 (either 10 mg/dose or 20 mg/dose) or 5 μg/kg/dose filgrastim used up to two weeks or stopped while ANC more than 5 × 109/L.

To track ANC concentration post chemotherapy, subjects returned to their study site for blood draws either daily (Cycle 1) or 3 times per week (every other day; Cycles 2-4) until ANC levels reached ≥2.0 × 109/L, post-nadir, and then every 3 days until the next chemotherapy cycle.

All subjects returned for an End of Study visit approximately 3 weeks after their final study drug administration (Study Day 84) and had a follow-up phone call 30 days after the last study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent and to compliant study procedure.
2. 18-70 years old;
3. Female with breast cancer patients after resection who planned to receive up to 4 cycles of chemotherapy (epirubicin and cyclophosphamide, 100 mg/m2 and 600 mg/m2, respectively).
4. Score 0-2 of East Cooperative Oncology Group (ECOG).
5. Absolute neutrophil count (ANC) ≥ 2.0 × 109/L, hemoglobin (Hb) ≥ 11.0 g/dl, and platelets (PLT) ≥ 100 × 109/L prior to chemotherapy.
6. Liver and kidney function tests were within normal range.
7. Left ventricular ejection fraction (LVEF) > 50%.
8. If female, subject is either not of childbearing potential, or is of childbearing potential.

Exclusion Criteria:

1. Patients received radiotherapy within 4 weeks prior to enrollment.
2. Patients received neoadjuvant chemotherapy prior to the resection for breast cancer.
3. Patients received bone marrow or hemopoietic stem cell transplantation.
4. Patient was with malignancy other than breast cancer.
5. Patients received G-CSF treatment within 6 weeks prior to enrollment.
6. Acute congestive heart failure, myocardial disease, or myocardial infarction diagnosed by clinical, electrocardiography, or any other medical procedure.
7. Any disease that possibly cause splenomegaly.
8. Acute infections, chronic active hepatitis B infection within 1 year (except subject with negative hepatitis B antigen prior to enrollment) or history of hepatitis C infection.
9. Pregnancy or lactating women; female with pregnancy potential had positive pregnancy test prior to study treatment.
10. Known the positive result of human immunodeficiency virus (HIV) or patients with acquired immune deficiency syndrome (AIDS).
11. Patients with active tuberculosis (TB), or had ever the history of close contact with patients with TB except negative result in tuberculin test; or under TB treatment; or suspected TB by chest X-ray.
12. Patients with sickle-cell anemia.
13. Patients with alcohol abuse or drug addiction that may affect the compliance of the study.
14. Patients with allergy to proteins extracted from Escherichia coli, G-CSF, or drug excipient.
15. Patients took other investigational products within 1 month or 5 half-lives prior to the enrollment (longer time period is preferred) based on the mechanism of action.
16. Patients with diseases or symptoms that may not be suitable to be enrolled in this study based on investigator's judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2015-09-20 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
The duration of moderate or severe (grade 3 and 4, respectively) neutropenia | In first of 4 cycles (21 days for each cycle) 84 days
  The duration of moderate or severe (grade 3 and 4, respectively) neutropenia post chemotherapy as measure of efficacy of F-627 compared to Filgrastim in female patients wiht breast cance receiving adjuvant chemotherapy.

SECONDARY OUTCOMES:
The incidence rates of Grade 3 and Grade 4 neutropenia | up to 4 cycles (84 days)
  The incidence rates of Grade 3 and Grade 4 neutropenia (ANC < 1.0 × 109/L and < 0.5 × 109/L, respectively) for all chemotherapy cycles.
The duration in days of Grade 3 and Grade 4 neutropenia for cycle 2 to 4. | cycle 2-4 (63 days)
  The duration in days of Grade 3 and Grade 4 neutropenia (ANC <1.0 × 109/L and ANC <0.5 × 109/L, respectively) for cycle 2 to 4.
The incidence rates of febrile neutropenia | Up to 4 cycles (84 days)
  The incidence rates of febrile neutropenia (FN; defined as a decrease in neutrophils associated with fever) for each chemotherapy cycle.
The depth of the ANC nadir | Up to 4 cycles (84 days)
  The depth of the ANC nadir for chemotherapy Cycles 1 to 4.
Number of participants with adverse events, changes from baseline of laboratory | Up to 4 cycles (84 days)
  Number of participants with adverse events, changes from baseline of laboratory values as measure of safety of F-627 compared to Filgrastim in female patients with breast cancer receiving chemotherapy.

OTHER OUTCOMES:
Immunogenicity of F-627 | Up to 4 cycles (84 days)
  Immunogenicity of F-627 by serum F-627 antibody analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Ji D, Wang S, Yao W, Hou D, Wang X, Ye C, Li H, Yang H, Yi J, Lu J, Wang H, Xu X, Cai D, Liu X, Yan X, Nie J, Cui S, Jiang H, Cao J. Efbemalenograstim Alfa, an Fc Fusion Protein, Long-Acting Granulocyte Colony-Stimulating Factor for Reducing the Risk of Chemotherapy-Induced Neutropenia: Results of a Phase II Randomized, Multicenter, Open-Label Trial. Clin Drug Investig. 2025 Nov;45(11):889-899. doi: 10.1007/s40261-025-01479-y. Epub 2025 Oct 9. PMID 41066031